CLINICAL TRIAL: NCT05418829
Title: An Open-Label Study to Evaluate the Long-Term Safety and Pharmacodynamic Efficacy of AT-007 in Adult Subjects With Classic Galactosemia (CG)
Brief Title: AT-007 in Adult Subjects With Classic Galactosemia (CG)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Applied Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-007-1006
Record Dates: First submitted 2022-02-16; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Classic Galactosemia
MeSH Terms: conditions — Galactosemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AT-007 (Experimental): Open-label AT-007 20 mg/kg once daily
  Interventions: Drug: AT-007

INTERVENTIONS:
Drug: AT-007 — AT-007 20 mg/kg once daily

SUMMARY:
This study is a 12-month open-label extension (OLE) study of AT-007 in adult subjects with CG who previously participated in Study AT-007-1001 Part D and/or Part D Extension.

The study is designed to assess the long-term safety of AT-007 in subjects with CG as well as the pharmacodynamics (PD) (inhibition of galactitol) and PK of AT-007. The effect of 12-month treatment with AT-007 on the levels of galactose and other galactose metabolites in subjects with CG will also be evaluated.

DETAILED DESCRIPTION:
Primary:

- To evaluate the long-term safety of 12-month oral administration of AT-007 in adult subjects with Classic Galactosemia (CG)

Secondary:

* To evaluate the long-term inhibition of galactitol, a biomarker of aldose reductase (AR) activity, induced by 12-month oral administration of AT-007 to adult subjects with CG
* To evaluate the pharmacokinetic (PK) parameters of 12-month oral administration of AT-007 in adult subjects with CG

Exploratory:

* To evaluate the effect of 12-month oral administration of AT-007 on the levels of galactose and its other metabolites in adult subjects with CG
* To evaluate the burden of illness (BOI) of adult subjects with CG
* To evaluate quality of life (QOL) measures of adult subjects with CG
* To evaluate the effect of 12-month oral administration of AT-007 on the BOI and QOL of adult subjects with CG

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female subject with a CG diagnosis
* Previous participation in Study AT-007-1001 Part D and/or Part D Extension
* No other significant health problems which preclude participation

Exclusion Criteria:

* Concomitant use of certain medications or over-the-counter therapies
* Discontinuation from Study AT-007-1001 Part D and/or Part D Extension due an adverse event

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety of 12-month oral administration of AT-007 in adult subjects with CG as assessed by adverse events. | 12 months
  Number of participants with treatment-emergent adverse events and broken down by organ class and relatedness.
To evaluate the long-term safety of 12-month oral administration of AT-007 in adult subjects with CG as assessed by clinical laboratory test results. | 12 months
  Number of participants with clinically-significant changes in clinical laboratory test results.
To evaluate the long-term safety of 12-month oral administration of AT-007 in adult subjects with CG as assessed by physical exam parameters. | 12 months
  Number of participants with clinically-significant changes in physical examination findings, vital sign abnormalities, and electrocardiogram findings.

SECONDARY OUTCOMES:
To evaluate the long-term change of galactitol, a biomarker of AR activity, induced by 12-month oral administration of AT-007 to adult subjects with CG | 12 months
To evaluate the pharmacokinetic (PK) parameter maximum concentration (Cmax) of 12-month oral administration of AT-007 in adult subjects with CG | 12 months
  Maximum concentration will be determined by individual concentration time-data (mg/L)
To evaluate the pharmacokinetic (PK) parameter Area-Under-the-Curve (AUC) of 12-month oral administration of AT-007 in adult subjects with CG (mg*h/L) | 12 months

OTHER OUTCOMES:
To evaluate the effect of 12-month oral administration of AT-007 on the levels of galactose and its other metabolites in adult subjects with CG | 12 months
To evaluate the burden of illness (BOI) of adult subjects with CG- Medical History | 12 months
  Narrative description of natural course of CG as extracted by chart review and physical exam findings noted in chart review including the baseline neurologic exam upon entering the clinical trial. (There are no units for a descriptive narrative of medical history)
To evaluate the burden of illness (BOI) of adult subjects with CG- NIH Motor Battery | 12 months
  NIH Motor Battery produces normalized percentile scores with higher scores being more normal. As an exploratory endpoint, changes in the score from baseline to month 12 will assessed.
To evaluate the burden of illness (BOI) of adult subjects with CG- Spiral Drawing Test | 12 months
  Spiral Drawing Test produces normalized percentile scores with higher scores being more normal. As an exploratory endpoint, changes in the score from baseline to month 12 will assessed.
To evaluate quality of life (QOL) measures of adult subjects with CG- PROMIS Emotional Distress questionnaire | 12 months
  The questionnaire assesses this function with higher scores relating to better function and may be used to compare over time for change from baseline to month 12. [PROMIS: Patient Reported Outcome Measure Information System]
To evaluate quality of life (QOL) measures of adult subjects with CG- PROMIS Emotional Support questionnaire | 12 months
  The questionnaire assesses this function with higher scores relating to better function and may be used to compare over time for change from baseline to month 12. [PROMIS: Patient Reported Outcome Measure Information System]
To evaluate quality of life (QOL) measures of adult subjects with CG- PROMIS Companionship questionnaire | 12 months
  The questionnaire assesses this function with higher scores relating to better function and may be used to compare over time for change from baseline to month 12. [PROMIS: Patient Reported Outcome Measure Information System]
To evaluate quality of life (QOL) measures of adult subjects with CG- PROMIS Social Isolation questionnaire | 12 months
  The questionnaire assesses this function with higher scores relating to better function and may be used to compare over time for change from baseline to month 12. [PROMIS: Patient Reported Outcome Measure Information System]
To evaluate quality of life (QOL) measures of adult subjects with CG- PROMIS Ability to Participate in Social Roles and Activities questionnaire | 12 months
  The questionnaire assesses this function with higher scores relating to better function and may be used to compare over time for change from baseline to month 12. [PROMIS: Patient Reported Outcome Measure Information System]

CONTACTS AND LOCATIONS:
Locations (1):
- Hassman Research Institute, Berlin, New Jersey, United States